CLINICAL TRIAL: NCT04871256
Title: Effects of Septorhinoplasty on Allergic Rhinitis Evolution
Brief Title: Effects of Septorhinoplasty on Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Pérez Sayáns (Other)
Collaborators: Universidade da Coruña (Other)
Responsible Party: Sponsor-Investigator, Mario Pérez Sayáns, Proffessor, University of Santiago de Compostela
Organization: University of Santiago de Compostela (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR/STP-UDC
Record Dates: First submitted 2021-01-14; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Allergic Rhinitis
Keywords: Septoplasty; VAS; quality of life; allergic rhinitis; nasal obstruction
MeSH Terms: conditions — Rhinitis, Allergic; Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: A prospective study with 1 months period follow up. Patients with septal deviation and allergic rhinitis diagnosis will be included. Obstruction airflow will be evaluated before and after surgery with rhinomanometry (RNM). Life quality will be assessed with VAS and ESPRINTquestionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inver (Experimental): Intervention: after screening, patient´s obstruction will be evaluated by anterior rhinomanometry (RNMa), and quality of life wil be scored through ESPRINT scale. ESPRINT is a validated Spanish questionnaire about daily life activity, sleep, psychology and perception of affection by allergic rhinitis.
  Symptoms will be evaluated with visual analogue scale (VAS) and clinical history. Symptoms like sneezing, itchy nose, ocular symptoms and/or nasal obstruction. Also medication (intranasal corticosteroid, antileukotrienes, antihistamine eye drops, antihistamine) frequency use will be registered
  Interventions: Procedure: Septorhinoplasty

INTERVENTIONS:
Procedure: Septorhinoplasty — This intervention will be performed by the same surgeon, after signing of patient inform consent.

SUMMARY:
Allergic rhinitis (AR) is a chronic inflammatory disease that affects almost 30% of adult population. Some patients associate septal deviation, main cause of chronic nasal obstruction, and AR. Current literature about AR treatment with septoplasty (STP) is still contradictory, because is thought that patients with AR are not able to appreciate improvement after surgery.

Patients diagnosed with allergic rinitis and septal deviation were evaluated to determined life quality and airflow obstruction evolution after STP.

DETAILED DESCRIPTION:
This is a prospective quasi experimental study. After being informed about the study, patients that signed written informed consent were included in the study. In week 0 before surgery, all measurements and questionnaires were performed. 1 month after surgery, measurements were repeated.

After screening, patient´s obstruction was evaluated by anterior rhinomanometry (RNMa), and quality of life scored through ESPRINT scale. ESPRINT is a validated Spanish questionnaire about daily life activity, sleep, psycology and perception of affection by allergic rhinitis. Symtoms were evaluated with visual analogue scale (VAS) and clinical history. Symptoms like sneezing, itchy nose, ocular symptoms and/or nasal obstruction. Also medication (intranasal corticosteroid, antileucotrienos, antihistamines eye drops , antishistamines) frequency use was registered.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Allergic Rhinitis
* Diagnosis of nasal obstruction with septal deviation

Exclusion Criteria:

* Previous nasal surgery
* Smokers
* Chronic obstructive pulmonary disease
* Psychiatric disorders
* Malignant tumors
* Severe hepatopathy
* Obstructive sleep apnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of Airflow rate | Change from baseline airflow rate (Before treatment) at 1 month after surgery
  Rhinomanometre will be used to determine airflow rate changes before surgery (septoplasty) and after it. Rhinomanometre will determine airflow rate in cm3/s and also use a quality scale as normal, mild, severe and very severe

SECONDARY OUTCOMES:
Changes from baseline of symptoms | Changes from baseline (Before treatment) at 1 month after surgery
  VAS score. VAS: visual analogue scale. Patients determine their symptoms with a visual scale that range from 0-10.
Changes from baseline in quality of life | Changes from baseline (Before treatment) at 1 month after surgery
  ESPRINT questionnaire. This is a validated spanish questionnaire about daily life impairments with 28 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Pérez Sayáns, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
Results will be shared by articles publication.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT04871256/Prot_SAP_ICF_000.pdf